CLINICAL TRIAL: NCT00251992
Title: Supportive Test for Acid-Related Symptoms (STARS II) With Esomeprazole and a Following 7-week, Double-blind, Randomized, Placebo Controlled Treatment Period in Uninvestigated Subjects With Upper Gastrointestinal Symptoms.
Brief Title: Nexium Dyspepsia/AST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SD-NED-0022; D9610C00022
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Gastrointestinal Disease; Signs and Symptoms, Digestive; Dyspepsia
MeSH Terms: conditions — Gastrointestinal Diseases; Signs and Symptoms, Digestive; Dyspepsia | interventions — Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole

SUMMARY:
The aim is to evaluate if the resolution of upper abdominal symptoms (pain or burning) during an acid suppressive test trial of esomprazole given daily for 7 days predicts symptoms resolution at the end of a subsequent treatment period of 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 months of symptoms of pain or burning centered in the upper abdomen prior to enrollment.
* Helicobacter pylori test performed at enrollment must be negative (Helicobacter pylori is a bacterial infection of the stomach).

Exclusion Criteria:

* Patients with symptoms of other gastrointestinal diseases, such as Gastroesophageal Reflux Disease (GERD), Irritable Bowel Syndrome (IBS) or Inflammatory Bowel Disease (IBD).
* Helicobacter pylori eradication treatment during the last 12 months prior to enrollment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1200
Dates: Start 2002-12; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome is whether the patient is a responder or not after 8 weeks treatment.
The primary efficacy outcome is based on symptom score recorded daily during the study in a patient diary.
The patient will judge their symptoms of pain or burning centered in the upper abdomen on a four-graded scale (none, mild, moderate or severe).

SECONDARY OUTCOMES:
The secondary efficacy outcomes are whether the patient is a responder or not after 4 weeks,
The average symptom score and the percentage of symptom-free days during the 7-week treatment period,
Presence/absence of specific GI symptoms after 4 and 8 weeks of therapy

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Nexium Medical Sciences Director, MD, Study Director — AstraZeneca
Locations (183):
- Austria (10):
  - Research Site, Braunau am Inn
  - Research Site, Graz
  - Research Site, Krems
  - Research Site, Linz
  - Research Site, Saint Johann
  - Research Site, Salzburg
  - Research Site, Sankt Pölten
  - Research Site, Vienna
  - Research Site, Wiener Neustadt
  - Research Site, Zell am See
- Belgium (21):
  - Research Site, Ans
  - Research Site, Brussels (Uccle)
  - Research Site, Gozée
  - Research Site, Halle
  - Research Site, Kontich
  - Research Site, Kortenberg
  - Research Site, Kraainem
  - Research Site, Liège
  - Research Site, Linkebeek
  - Research Site, Massemen
  - Research Site, Moerkerke
  - Research Site, Natoye
  - Research Site, Oud-Heverlee
  - Research Site, Saint-Médard
  - Research Site, Soignies
  - Research Site, Waremme
  - Research Site, Wezembeek-Oppem
  - Research Site, Wingene
  - Research Site, Zoersel
  - Research Site, Zolder
  - Research Site, Zonhoven
- Canada (39):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, Penticton, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Bay Roberts, Newfoundland and Labrador
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Elmsdale, Nova Scotia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Ajax, Ontario
  - Research Site, Brampton, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Dorchester, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Kanata, Ontario
  - Research Site, Kitchener, Ontario
  - Research Site, London, Ontario
  - Research Site, Markham, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Niagara Falls, Ontario
  - Research Site, North York, Ontario
  - Research Site, Orléans, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Richmond Hill, Ontario
  - Research Site, Saint Catherines, Ontario
  - Research Site, Sainte Gedeon-de-Beauce, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Stirling, Ontario
  - Research Site, Thunder Bay, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Tottenham, Ontario
  - Research Site, Whitby, Ontario
  - Research Site, Charlottetown, Prince Edward Island
  - Research Site, Parkdale, Prince Edward Island
  - Research Site, Charlesbourg, Quebec
  - Research Site, Granby, Quebec
  - Research Site, Saint-Léonard, Quebec
  - Research Site, Sainte-Foy, Quebec
- Finland (9):
  - Research Site, Espoo
  - Research Site, Helsinki
  - Research Site, Kouvola
  - Research Site, Lempäälä
  - Research Site, Pirkkala
  - Research Site, Pori
  - Research Site, Sahalahti
  - Research Site, Tampere
  - Research Site, Vääksy
- France (10):
  - Research Site, Angers
  - Research Site, Dambach-la-Ville
  - Research Site, Dijon
  - Research Site, La Seyne-sur-Mer
  - Research Site, Laxou
  - Research Site, Louviers
  - Research Site, Mont-de-Marsan
  - Research Site, Nancy
  - Research Site, Saint-Ouen
  - Research Site, Vieux-Condé
- Germany (3):
  - Research Site, Lochham
  - Research Site, München
  - Research Site, Rödental
- Hungary (8):
  - Research Site, Budaörs
  - Research Site, Budapest
  - Research Site, Esztergom
  - Research Site, Hatvan
  - Research Site, Nagykanizsa
  - Research Site, Siófok
  - Research Site, Tát
  - Research Site, Zalaegerszeg
- Mexico (6):
  - Research Site, México, D.F
  - Research Site, Culiacán
  - Research Site, Guadalajara
  - Research Site, León
  - Research Site, México
  - Research Site, Torreón
- Norway (15):
  - Research Site, Bekkestua
  - Research Site, Bergen
  - Research Site, Hønefoss
  - Research Site, Lier
  - Research Site, Lysaker
  - Research Site, Moss
  - Research Site, Oslo
  - Research Site, Paradis
  - Research Site, Rådal
  - Research Site, Rykkin
  - Research Site, Sandefjord
  - Research Site, Skien
  - Research Site, Søgne
  - Research Site, Tvedestrand
  - Research Site, Østerås
- South Africa (8):
  - Research Site, Lenasia, Gauteng
  - Research Site, Bloemfontein
  - Research Site, Boksburg
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Halfway House
  - Research Site, Lyttelton Manor
  - Research Site, Pretoria
- Sweden (24):
  - Research Site, Ängelholm
  - Research Site, Fritsla
  - Research Site, Gothenburg
  - Research Site, Halmstad
  - Research Site, Höganäs
  - Research Site, Ingelstad
  - Research Site, Jönköping
  - Research Site, Kalmar
  - Research Site, Kilafors
  - Research Site, Kristinehamn
  - Research Site, Kungsör
  - Research Site, Motala
  - Research Site, Munkedal
  - Research Site, Nässjö
  - Research Site, Norrtälje
  - Research Site, Rättvik
  - Research Site, Staffanstorp
  - Research Site, Sundsbruk
  - Research Site, Trollhättan
  - Research Site, Uddevalla
  - Research Site, Upplands Vasby
  - Research Site, Vaxjo
  - Research Site, Vällingby
  - Research Site, Västerås
- Switzerland (9):
  - Research Site, Schönbühl-Urtenen, Canton of Bern
  - Research Site, Egg Bei Zürich, Canton of Zurich
  - Research Site, Winterthur, Canton of Zurich
  - Research Site, Zurich, Canton of Zurich
  - Research Site, Aarau
  - Research Site, Brittnau
  - Research Site, Küttigen
  - Research Site, Schaffhausen
  - Research Site, Zurich
- United Kingdom (21):
  - Research Site, Ely, Cambridgeshire
  - Research Site, Woking, Surrey
  - Research Site, Audley
  - Research Site, Blackburn
  - Research Site, Blackpool
  - Research Site, Chesterfield
  - Research Site, Coventry
  - Research Site, Enfield
  - Research Site, Glasgow
  - Research Site, Hadleigh
  - Research Site, Harrow
  - Research Site, Irvine
  - Research Site, Mansfield
  - Research Site, Nottingham
  - Research Site, Royal Tunbridge Wells
  - Research Site, Sheffield
  - Research Site, Shrewsbury
  - Research Site, Slough
  - Research Site, Titchfield
  - Research Site, Tonbridge
  - Research Site, Watford

REFERENCES:
- [Derived] van Zanten SV, Wahlqvist P, Talley NJ, Halling K, Vakil N, Lauritsen K, Flook N, Persson T, Bolling-Sternevald E; STARS II Investigators. Randomised clinical trial: the burden of illness of uninvestigated dyspepsia before and after treatment with esomeprazole--results from the STARS II study. Aliment Pharmacol Ther. 2011 Oct;34(7):714-23. doi: 10.1111/j.1365-2036.2011.04789.x. Epub 2011 Aug 17. PMID 21848799
- [Derived] van Zanten SV, Flook N, Talley NJ, Vakil N, Lauritsen K, Bolling-Sternevald E, Persson T, Bjorck E, Svedberg LE; STARS II Study Group. One-week acid suppression trial in uninvestigated dyspepsia patients with epigastric pain or burning to predict response to 8 weeks' treatment with esomeprazole: a randomized, placebo-controlled study. Aliment Pharmacol Ther. 2007 Sep 1;26(5):665-72. doi: 10.1111/j.1365-2036.2007.03409.x. PMID 17697200